CLINICAL TRIAL: NCT02527382
Title: Peritoneal Bacterial Contamination With Closed or Open Rectal Stump
Brief Title: Peritoneal Bacterial Contamination Following Resection With Closed or Open Rectal Stump for Left-sided Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florin Iordache (Other)
Responsible Party: Sponsor-Investigator, Florin Iordache, Senior Lecturer of General Surgery, Attending Surgeon, Bucharest Emergency Hospital
Organization: Bucharest Emergency Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 23937
Record Dates: First submitted 2015-08-16; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Bacterium-Related Malignant Neoplasm

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Closed stump (Experimental): Before cutting the bowel, a peritoneal sample for bacterial culture is taken from the peritoneal cavity (pelvic pouch). Anastomosis is performed while a distal clamp is placed on the rectal stump.
  Interventions: Procedure: Closed stump
- Open stump (No Intervention): Before cutting the bowel, a peritoneal sample for bacterial culture is taken from the peritoneal cavity (pelvic pouch). Anastomosis is performed while no distal clamp is placed on the rectal stump.

INTERVENTIONS:
Procedure: Closed stump — Before cutting the bowel, a peritoneal sample for bacterial culture is taken from the peritoneal cavity (pelvic pouch). Anastomosis is performed while a bowel clamp is placed on the rectal stump. A second bacterial sample is obtained at the completion of the anastomosis from the same place (pelvic pouch) as the first one.
  Arms: Closed stump

SUMMARY:
The purpose of this study is to check if there is a difference in peritoneal contamination in patients undergoing rectal resection with closed and open rectal stump prior to anastomosing.

DETAILED DESCRIPTION:
There is not much information regarding the peritoneal bacterial contamination during colorectal surgery. The null hypothesis is that there is no difference in peritoneal contamination following resection with closed or open rectal stump for left-sided cancer. Patients scheduled for elective resection are allocated for open resection with the distal stump closed or open. Anastomosis is performed while a clamp is placed on the rectal stump in one arm of the study while in the other arm, the stump remains open until the anastomosis is completed. A second bacterial sample will be obtained at the completion of the anastomosis from the same place (pelvic pouch) as the first one. After sampling an air leak test will be performed. A quantitative assessment of the number of Colony Forming Units (CFU/ml) of aerobic and anaerobic bacteria will be done for each patient. Operative time and time interval between samples will be measured. Postoperatively, possible complications (surgical site infections, leakage) will be monitored. The primary objective will be to determine the differences in peritoneal contamination between closed and open rectal stump during colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult patients scheduled for a left colectomy, sigmoidectomy or rectal resection with a proposed anastomosis at the level of the rectum agreeing to participate in the study.

Exclusion Criteria:

* Patients without informed consent
* Class V patients on American Society of Anesthesiologists (ASA) of Physical Health Score
* Patient with prior peritonitis
* Patients with acute inflammatory bowel disease
* Recent antibiotic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The number of Colony-Forming Units (CFU)/ml from the peritoneal samples | within the first 30 days after surgery
  The formula we will use is: number of CFU (colony forming units)/ml = n x 10 x d, where n = number of colonies on the media and d = dilution reverse. The final number of CFU/ml will be given as the arithmetic mean of the three dilutions done for each sample. When no bacterial growth is found the results are given as 0 CFU/ml. The maximum limit is considered 100,000 CFU/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Florin M Iordache, MD, Principal Investigator — Bucharest Emergency Hospital